CLINICAL TRIAL: NCT06840119
Title: A Phase 1/2 First-in-Human Study of the Safety and Efficacy of IMC-R117C (PIWIL1 × CD3 ImmTAC® Bispecific Protein) as a Single Agent and in Combination in HLA-A*02:01-Positive Participants With Selected Advanced PIWIL1-Positive Cancers
Brief Title: Phase 1/2 Study of IMC-R117C in Selected Advanced Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immunocore Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMC-R117C-1004; 2023-508090-87-00 (Other: EU CTR)
Record Dates: First submitted 2025-02-05; First posted 2025-02-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cancer; HLA-A*02:01-positive
MeSH Terms: conditions — Neoplasms | interventions — Angiogenesis Inhibitors; Antibodies, Monoclonal

STUDY DESIGN:
Intervention Model Description: The study will include sequential assignment for non-randomized and randomized arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A: IMC-R117C Monotherapy Dose-Escalation (Experimental): Participants receive IMC-R117C intravenous (IV) infusion.
  Interventions: Drug: IMC-R117C
- Arm B: IMC-R117C Combination Dose-Escalation (Experimental): Participants receive IMC-R117C IV infusion in combination with standard of care chemotherapy and antiangiogenic agent
  Interventions: Drug: IMC-R117C; Drug: Chemotherapy drug; Drug: Antiangiogenic Agent
- Arm C: IMC-R117C Combination Dose-Escalation (Experimental): Participants receive IMC-R117C IV infusion with targeted therapies
  Interventions: Drug: IMC-R117C; Drug: Kinase inhibitor; Drug: Monoclonal antibody
- Arm D: Control Arm (Active Comparator): Participants receive standard of care chemotherapy and antiangiogenic agent
  Interventions: Drug: Chemotherapy drug; Drug: Antiangiogenic Agent

INTERVENTIONS:
Drug: IMC-R117C — IV infusion
  Arms: Arm A: IMC-R117C Monotherapy Dose-Escalation; Arm B: IMC-R117C Combination Dose-Escalation; Arm C: IMC-R117C Combination Dose-Escalation
Drug: Chemotherapy drug — IV infusion
  Arms: Arm B: IMC-R117C Combination Dose-Escalation; Arm D: Control Arm
Drug: Chemotherapy drug — oral
  Arms: Arm B: IMC-R117C Combination Dose-Escalation
Drug: Kinase inhibitor — oral
  Arms: Arm C: IMC-R117C Combination Dose-Escalation
Drug: Antiangiogenic Agent — IV infusion
  Arms: Arm B: IMC-R117C Combination Dose-Escalation; Arm D: Control Arm
Drug: Monoclonal antibody — IV infusion
  Arms: Arm C: IMC-R117C Combination Dose-Escalation

SUMMARY:
This phase 1/2 first-in-human study is designed to test the safety and efficacy of IMC-R117C (PIWIL1 × CD3 ImmTAC® Bispecific Protein) as a single agent and in combination with other therapies in HLA-A*02:01-positive participants with selected advanced PIWIL1-Positive cancers.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* HLA-A*02:01-positive
* Histologically confirmed advanced colorectal, esophageal, gastric, or ovarian carcinoma
* Archived or fresh tumor tissue sample that must be confirmed as adequate
* Evaluable/Measurable disease per RECIST 1.1
* Previously received applicable standard treatments
* Male and female participants of childbearing potential who are sexually active with a non-sterilized partner must agree to use highly effective methods of birth control

Exclusion Criteria:

* Symptomatic or untreated central nervous system metastasis
* Recent bowel obstruction
* Ongoing ascites or effusion requiring recent drainages
* Significant ongoing toxicity from prior anticancer treatment
* Out-of-range laboratory values
* Clinically significant lung, heart, or autoimmune disease
* Ongoing requirement for immunosuppressive treatment
* Significant secondary malignancy
* Hypersensitivity to study drug or excipients
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Percentage of participants with ≥1 dose-limiting toxicity (DLT) | Up to ~24 months
Dose Escalation: Percentage of participants with ≥1 adverse event (AE) | Up to ~24 months
Dose Escalation: Percentage of participants with ≥1 serious adverse event (SAE) | Up to ~24 months
Dose Escalation: Percentage of participants with significant changes in electrocardiogram (ECG) recordings | Up to ~24 months
Dose Escalation: Percentage of participants with significant changes in vital signs | Up to ~24 months
Dose Escalation: Percentage of participants with significant changes in laboratory results | Up to ~24 months
Dose Escalation: Percentage of participants with a dose interruption, reduction, or discontinuation | Up to ~24 months
Expansion: Best Overall Response (BOR) as Determined by RECIST v1.1 | Up to ~24 months

SECONDARY OUTCOMES:
Dose Escalation: Best Overall Response (BOR) as Determined by RECIST v1.1 with IMC-R117C Monotherapy and in Combination | Up to ~36 months
Dose Escalation: Duration of Response (DOR) as Determined by RECIST v1.1 with IMC-R117C Monotherapy and in Combination | Up to ~36 months
Dose Escalation: Progression-free survival (PFS) as Determined by RECIST v1.1 with IMC-R117C Monotherapy and in Combination | Up to ~36 months
Dose Escalation: Overall Survival (OS) with IMC-R117C Monotherapy and in Combination | Up to ~36 months
Expansion: Duration of Response (DOR) as Determined by RECIST v1.1 with IMC-R117C Monotherapy | Up to ~36 months
Expansion: Progression-free survival (PFS) as Determined by RECIST v1.1 with IMC-R117C Monotherapy | Up to ~36 months
Expansion: Overall Survival (OS) with IMC-R117C Monotherapy | Up to ~36 months
Expansion: Percentage of participants with ≥1 Adverse Events (AE) | Up to ~24 months
Expansion: Percentage of participants with ≥1 Serious Adverse Events (SAE) | Up to ~24 months
Expansion: Percentage of participants with significant changes in electrocardiogram (ECG) recordings | Up to ~24 months
Expansion: Percentage of participants with significant changes in vital signs | Up to ~24 months
Expansion: Percentage of participants with significant changes in laboratory findings | Up to ~24 months
Expansion: Percentage of participants with dose interruptions, reductions, or discontinuation | Up to ~24 months
All Study: Plasma Concentration of IMC-R117C | Up to ~36 months
All Study: Incidence of anti-IMC-R117C Antibody Formation | Up to ~36 months
All Study: Incidence of tumor expression and localization of PIWIL1 | Up to ~36 months

CONTACTS AND LOCATIONS:
Locations (13):
- Australia (2):
  - St Vincent's Hospital, Darlinghurst, Sydney
  - Peter MacCallum Cancer Centre, Melbourne
- Belgium (3):
  - Institut Jules Bordet, Anderlecht
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Universitaetsklinikum Heidelberg, Heidelberg, Germany
- Italy (2):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - nstituto Clinico Humanitas, Rozzano
- Antoni van Leeuwenhoek, Amsterdam, Netherlands
- Spain (4):
  - Hospital HM Nou Delfos, Barcelona
  - VHIO, Vall d'Hebron University Hospital, Barcelona
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid